CLINICAL TRIAL: NCT01189825
Title: Effects of Acute Exercise on Sexual Arousal in Women Taking a Selective Serotonin Reuptake Inhibitor (SSRI) or Selective Serotonin/Norepinephrine Reuptake Inhibitor
Brief Title: Efficacy of Exercise for Sexual Side Effects of Antidepressants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Tierney Kyle Ahrold Lorenz, Researcher, University of Texas at Austin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2007-12-0059; 1F31MH085416-01A1 (NIH)
Record Dates: First submitted 2010-08-25; First posted 2010-08-27 (Estimated); Last update posted 2013-02-27 (Estimated); Status verified 2013-02

CONDITIONS: Sexual Dysfunction
Keywords: Physiological; Antidepressive Agents
MeSH Terms: conditions — Sexual Dysfunction, Physiological | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exercise (Experimental)
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Moderate to intense cardiovascular exercise on a treadmill for 20 minutes

SUMMARY:
The major aim of the this study is to replicate findings of previous research that examined the effects of acute exercise on sexual arousal in women in a novel population, namely, women taking antidepressants of the selective serotonin reuptake inhibitors (SSRI) or selective serotonin and norepinephrine reuptake inhibitors (SNRI) class. In previous studies it has been found that acute, moderate-intensity exercise facilitated physiological sexual arousal responses in healthy, sexually functional women. However, it is known that antidepressants may induce sexual dysfunction, and thus in the present study, the investigators are examining whether acute exercise may facilitate sexual responses in women with taking antidepressants, including women with antidepressant-related sexual dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* female
* age 18 or older
* currently receiving a consistent dosage of escitalopram, citalopram, sertraline, desvenlafaxine, venlafaxine, or duloxetine
* currently sexually active
* willing and able to exercise
* experiencing regular menstrual cycles
* not currently pregnant and not intending to become pregnant during trial

Exclusion Criteria:

* currently taking more than one psychoactive medication
* factors indicating risk of cardiovascular activity, including acute or chronic cardiovascular illness, including clinically significant hypertension (defined as self-reported hypertension or "blood pressure greater than 140/90" or receiving medications designed to treat hypertension); recent chest pain; frequent or recurrent faint or dizzy spells; severe or untreated exercise-related asthma; or musculoskeletal illness or injury that would be expected to worsen with physical exercise. Additionally, women will be excluded if they are found to have any of the following as measured during the fitness assessment of the first session: a BMI over 40, waist circumference over 40 inches, waist-to-hip ratio of greater than 0.9, systolic blood pressure greater than 150 or diastolic pressure over 95, or resting heart rate over 90.
* factors associated with significant genital nerve damage, including: previous major pelvic surgery that may have caused nerve damage, including hysterectomy, vulvectomy, circumcision, colostomy, cystostomy, or serious bladder, rectal, or abdominal surgery; or neurological impairment due to diabetes, stroke, pelvic nerve damage secondary to trauma, cancer treatments, myasthenia gravis, multiple sclerosis or spinal cord damage.
* factors associated with non-normative endocrine function, including: perimenopausal or menopausal status, or >1 missed menstrual period in the previous 6 months; or currently pregnant, breastfeeding, or having breastfed within the past 3 months; or reporting clinically significant untreated renal or endocrine disease
* untreated serious mental health conditions
* sexual aversion or distress due to history of unwanted sexual contact

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2009-06; Primary Completion 2011-05 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Sexual arousal | 5 & 15 minutes post exercise
  Arousal to sexually explicit stimuli will be measured in the laboratory using a vaginal photoplethysmograph.

CONTACTS AND LOCATIONS:
Overall Officials: Tierney K Ahrold Lorenz, M.A., Principal Investigator — University of Texas at Austin
Locations (1):
- University of Texas at Austin, Austin, Texas, United States

REFERENCES:
- See also: Laboratory webpage — http://www.mestonlab.com